CLINICAL TRIAL: NCT03196128
Title: Digital Media Versus Standard Method of Communication to Examine Engagement of Patients in Community Early Intervention Psychosis (EIP) Services
Brief Title: Early Intervention Psychosis Communication and Engagement Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Christina Clark, Lead Investigator, South London and Maudsley NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17/EM/0093
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: First Episode Psychosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital (Active Comparator)
  Interventions: Other: Digital communication
- Non Digital (Active Comparator)
  Interventions: Other: Non digital

INTERVENTIONS:
Other: Digital communication — Communicating with patients via email and text message.
  Arms: Digital
Other: Non digital — Communicating with patients via telephone and written appointment letters.
  Arms: Non Digital

SUMMARY:
This study will examine whether or not the use of digital communication methods (text messages and emails) improves patient engagement with Early Intervention Psychosis (EIP) Services, compared to standard communication methods (letters and telephone calls).

One of the biggest challenges of psychiatric services is patient disengagement. People with psychosis, are often difficult to engage in community based mental health services (CMHTs). Patient's who disengage from psychiatric care often have higher social care needs, are often more unwell and are more likely to be detained under the Mental Health Act compared to those who engage. It is important to examine the reasons for this for both research and clinical reasons to establish the effectiveness of the service to its users. Importance must be placed on the clinician's perspective of the engagement; the patient's perspective is vital.

This study is a pilot two-arm pragmatic Randomised Control Trial to examine the feasibility of assessing engagement of EIP services through different communication methods. Patients and care-coordinators will use self-reported scales to measure engagement to determine whether this improves through the use of different communication methods.

Patients will be asked to consent to being randomly allocated to one of two groups:

(i.) Receive letters, phone calls and voicemail's from their care coordinator for standard appointments.

OR

(ii.) Receive text messages and emails from their care-coordinator for standard appointments.

Patients eligible for this study will be in their first six months of care under an EIP CMHT and who have consented to take part. They will be aged 18-35, not a hospital inpatient, have access to the Internet, a mobile phone and who are fluent in the English language.

Care-coordinators will assess the feasibility and acceptability of the design and procedures and determine an effective sample size calculation for a future large scale pragmatic Randomised Controlled Trial.

DETAILED DESCRIPTION:
Participants (patients and care-coordinators):

Instruments:

Patients:

SOLES (Singh O'Brien Level of Engagement Scale, O'Brien et al 2009). (Appendix 1) This self-reporting scale is designed to measure the level of engagement in people with psychosis. It contains 16 questions covering various aspects of engagement, each question scored in a scale ranging from 0-10. This scale takes about 8-10 minutes to be completed.

Care Coordinators:

SES (Service Engagement Scale, Tait et al 2002). (Appendix 2) The SES is a scale completed by clinicians to assess their perceived level of engagement of patients under their care. It is a 14-question scale covering the same areas as the SOLES. The scale taken about 4-6 minutes to be completed.

Care Coordinator Feasibility Questionnaire:

It would also be of interest to collect feedback from care coordinators about the ease of use of the procedure along with the relevance and acceptability. This will be done through the use of a self reporting scale of how feasible the intervention delivery was. (Appendix 3)

Interventions:

When arranging appointments or having any other communication outside face-to-face meetings, care coordinators participating in this study will be expected to contact their patients in two distinct ways:

(i) 20 patients will receive Standard contact: this will happen by means of letters, telephone call and voicemail's only. Care co-ordinators already have trust mobile phones that they can use.

(ii) 20 patients will receive Digital media contact: only text messages and e-mails will be used to contact patients. Care coordinators will also be provided with i-pads (funded by the British Research Council so that they can do this when also outside of clinic).

Both types of contact will be made explicit for care coordinators at the beginning of the study, with frequent reminders occurring during the period of data collection. Care coordinators will have immediate access to written information about each of the interventions through participant information and consent forms provided (appendix 5).

Design:

A two-arm pragmatic pilot Randomised Controlled Trial. will be conducted comparing the digital media contact methods with standard contact methods and will assess the potential for progressing into a full pragmatic Randomised Controlled Trial. The co-primary outcome measures are to determine whether engagement with care coordinator/services improves through the use of digital media communication compared to standard methods of communication using The Singh O'Brien Level of Engagement Scales (SOLES)(O'Brien et al 2009) (SOLES) and The Service Engagement Scale (SES) (Tait et al 2002). These are self rating scales which will be completed both pre and post intervention to examine whether or not there has been an increase in engagement. Success of the study will be measured by an increase of scores in the scales to determine whether or not increased engagement was achieved.

Procedures:

Consecutive patients accepted for care under EIP teams will be asked to consent to participate in this study. If they consent, they will be allocated to one of two groups: either the Standard group or the Digital Media group. It is expected that each group will have approximately 20 patients. Care coordinator's will also be asked to consent to participate in the study and will be briefed by chief investigator on procedures.

Two months after intake into the study, patients and care coordinators will complete their respective engagement questionnaires. The level of engagement of each group, as measured by the instruments, will be used to analyse and compare the impact of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* First Episode Psychosis under the care of Early Intervention Psychosis Team Community Mental Health Team.
* Aged 18 - 65
* Fluent in the English language
* In first six months of service
* Has a mobile phone and access to the internet/email

Exclusion Criteria:

* Currently an inpatient in hospital
* Nearing discharge from EIP services
* Is not fluent in the English Language
* In acute crisis at the time of participant recruitment
* Does not have a mobile phone or access to the internet/email

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2018-01-30 (Estimated)

PRIMARY OUTCOMES:
Singh O'Brien Level of Engagement Scale | Average completion time - 8-10 minutes.
  Self reporting scale designed to measure the level of engagement in people with psychosis. It contains 16 questions covering various aspects of engagement, each question scored in a scale ranging from 0-10.
Service Engagement Scale | Average completion time: 4- 6 minutes.
  A scale completed by clinicians to assess their perceived level of engagement of patients under their care. It is a 14 - question scale covering the same areas as the SOLES.

SECONDARY OUTCOMES:
Care Coordinator Feasibility Questionnaire | Average completion Time: 10 minutes.
  Self reporting scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Christina Clark, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No